CLINICAL TRIAL: NCT06280742
Title: Study of Neuroinflammation in Multiple Sclerosis by PET-MRI Imaging Using the Radiotracer ([18F]-DPA-714) : a Multicentre Cohort Study
Brief Title: Study of Neuroinflammation in Multiple Sclerosis by PET-MRI Imaging Using the Radiotracer ([18F]-DPA-714) : a Multicentre Cohort Study (INFLANET)
Acronym: INFLANET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP221366
Record Dates: First submitted 2024-01-23; First posted 2024-02-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; PET-MRI
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Experimental): MRI with added injection of gadolinium
  Interventions: Radiation: PET-MRI with [18F]-DPA-714
- Healthy Volunteers (Active Comparator)
  Interventions: Radiation: PET-MRI with [18F]-DPA-714

INTERVENTIONS:
Radiation: PET-MRI with [18F]-DPA-714 — PET-MRI with [18F]-DPA-714

SUMMARY:
The Service Hospitalier Frédéric-Joliot (SHFJ) and Paris Brain Institute (ICM) groups have identified [18F]-DPA-714 as a promising second-generation TSPO tracer, a macromolecule overexpressed in neuroinflammatory conditions, for PET imaging. They have also developed a non-invasive quantification methodology, enabling the generation of individual neuroinflammation maps in MS patients. Recent findings from [18F]-DPA-714 PET imaging in MS patients revealed that most of the white matter lesions contained a smoldering component, even when considered inactive on MRI, and that their neuroinflammatory profiles were associated with longitudinal disability worsening. The Inflanet project aims to leverage a unique consortium comprising French radiochemists, radiopharmacists, nuclear medicine/neuroimaging experts, and MS neurologists to establish the first national network dedicated to [18F]-DPA-714 PET imaging in MS, so far limited to monocentric studies.

The objectives of the INFLANET project are (1) to conduct the first multicenter study assessing neuroinflammation in patients with active MS using [18F]DPA-714 PET tracer, and (2) to establish a methodology suitable for the quantification of multicenter PET data obtained with [18F]DPA-714. The INFLANET initiative aims to disseminate TSPO PET within the French MS research community, thereby opening the unique perspective of future large-scale, multicenter studies. These endeavors are expected to enhance our capacity to predict diseases, stratify patients, and assess new therapeutic interventions.

DETAILED DESCRIPTION:
INFLANET is a multicentric, prospective, non-randomized, non-blinded, interventional study.The study will include a total of 41 participants, with 18 individuals diagnosed with multiple sclerosis (MS) distributed across three sites (6 patients per site: Paris, Lyon, Rennes). Additionally, there will be 23 healthy volunteers (HV), with 20 HV allocated to the Lyon and Rennes sites (10 HV per site) and 3 HV for the Paris site.

The study involves several clinical visits, with two visits for patients (Screening V0 and Baseline V1), two visits for 20 healthy volunteers (Screening V0 and Baseline V1), and three visits for three healthy volunteers (Screening V0, Baseline V1 - Test, and V1' - Retest, in Paris site). Various evaluations are integrated into the study, including neurological assessments at the screening visit, neuropsychological assessments at the baseline visit, 18F-DPA714 PET-MR or PET + MRI (n=1 for 20 HV and 18 subjetcs with MS; n=2 for 3 HV) at V1 and V1', and blood sampling at the screening visit to confirm TSPO eligibility.

The PET-MR procedure involves TSPO PET using [18F]-DPA-714 in conjunction with 3T MRI for both MS patients and healthy volunteers. Gadoteric acid is administered for MS patients only as part of the imaging.

ELIGIBILITY:
Inclusion Criteria:

RRMS patients:

* Age between 18 and 55 years old
* RRMS according to the 2017 Mc Donald criteria
* At least 9 supra-tentorial white matter lesions on T2/FLAIR MRI
* Last treatment with methylprednisolone should have been performed at least 1 month before PET examinations
* No current disease modifying therapy
* Indication for a highly active disease modifying treatment: Natalizumab, anti CD20 antibody, Alemtuzumab, sphingosine-1 phosphate modulator, or cladribine. This will consist either as patients with an active form of relapsing MS or patients who have experienced two relapses during the previous year
* Affiliation to a social security scheme or beneficiary of such a scheme (except "Aide Médicale d'Etat")

Healthy Volunteers:

* Age between 18 and 55 years old
* Without any evolutive pathology
* Able to understand the study objectives and procedures
* Affiliation to a social security scheme or beneficiary of such a scheme (except "Aide Médicale d'Etat")

Exclusion Criteria:

For all participants:

* Any reasons, which does not allow to perform MRI, including claustrophobia, the implant of a pace-maker or the presence of an intra-ocular foreign body, (a contra-indication questionnaire will be filled in beforehand)
* Realization of any test using radioactivity within the last 12 months
* Low Affinity Binding profile (analyse of TSPO polymorphism done at screening visit)
* Pregnancy, breast-feeding, lack of efficient contraception for women of childbearing potential
* Current symptoms of severe or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary or cardiac disease, or any other chronic neurological diseases
* Unwillingness to be informed in case of unexpected MRI abnormality (with a significant medical anomaly)
* Patient under legal protection
* Participation in another interventional study or being in the exclusion period at the end of a previous study

RRMS patients:

* Hypersensitivity to gadoteric acid
* Meglumine or any drug containing gadolinium
* Severe renal insufficiency (creatinine clearance < 60mL/min and GFR <30ml / min / 1.73m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To quantify the smoldering component of white matter lesions in people with MS, as compared with [18F]-DPA-714 binding in the white matter of HC who underwent a PET a acquisition with the same camera camera than patients in each center. | 26 month
  The respective proportion of lesions classified as homogeneously active, rim active and inactive for every single patient with MS. Classification of lesions will be based on predefined data-driven threshold of activity in lesions subareas (Hamzaoui et al, 2023).

SECONDARY OUTCOMES:
To quantify for each patient the regional neuroinflammatory load, measured as [18F]-DPA-714 DVR, in specific regions of interest: total brain, normal appearing white matter, cortex, thalami, deep grey matter. | 26 month
  Regional mean and voxel wise individual maps of innate immune cells activation derived from baseline [18F]-DPA-714 PET : they will be expressed as mean DVR values and as percentage of voxel classified as "DPA+", for each region of interest: whole brain, NAWM, grey matter, cortex, thalami, deep grey matter, white matter T2 lesions, white matter T1 lesions.
The MRI signatures of each lesional subtypes, and correlation between MRI metrics and [18F]-DPA-714 DVR in each region of interest. | 26 month
  MRI data: T1, T2, FLAIR, SWI, QSM, MTR, ihMT, diffusion collected at baseline. This will include the assessment of novel algorithms that have been generated through deep learning and attempt to reproduce PET using multimodal MRI datasets.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Département de Neurologie,Pierre Wertheimer Neurological Hospital, Lyon
  - CERMEP, Lyon
  - CIC Neurosciences, GH Pitié-Salpêtrière, Paris
  - Centre Eugène Marquis, Rennes
  - Service de Neurologie, CHU Pontchaillou, Rennes
  - CHU Toulouse - Département de Neurologie, Toulouse
  - CHU Toulouse - Service de médecine nucléaire, Toulouse

IPD SHARING:
Plan to Share IPD: No